CLINICAL TRIAL: NCT05035355
Title: A Spontaneous Breathing Trial-based Protocol-directed Program in Difficult-to-Wean Patients
Brief Title: A SBT-based Protocol-directed Program in Difficult-to-Wean Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: JinyanXing (Other)
Responsible Party: Sponsor-Investigator, JinyanXing, Director, The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QYFYWZLL26347
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Respiration, Artificial
Keywords: Protocol-directed weaning; Mechanical ventilation; High-flow nasal cannula; Spontaneous breathing trial
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- weaning protocol group (Experimental): spontaneous breathing trial (SBT)-based protocol-directed weaning combined with the high-flow nasal cannula group
  Interventions: Procedure: a weaning protocol
- routine SBT weaning group (No Intervention)

INTERVENTIONS:
Procedure: a weaning protocol — a weaning protocol that is combined spontaneous breathing trial (SBT) with the high-flow nasal cannula (HFNC)
  Arms: weaning protocol group

SUMMARY:
Weaning patients from a ventilator is one of the most challenging processes in an intensive care unit. The investigators aimed to determine whether spontaneous breathing trial (SBT)-based protocol-directed weaning combined with the high-flow nasal cannula (HFNC) could be superior to routine SBT-based weaning in reducing the duration of mechanical ventilation (MV) in difficult-to-wean patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 16 years old
* MV for more than 48 hours
* intubated or tracheostomized

Exclusion Criteria:

* pregnancy
* irreversible respiratory failure caused by neurodegenerative disorders, such as Alzheimer disease, motor neuron disease, or multiple system atrophy
* pre-existing decision to limit life support
* waiving of MV during treatment
* terminal stage of severe illness

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
mechanical ventilation days | 60 days
  the duration of mechanical ventilation

SECONDARY OUTCOMES:
re-intubated within 24 hours | 24 hours
  re-intubated within 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided